CLINICAL TRIAL: NCT02321423
Title: International Pachyonychia Congenita Research Registry
Acronym: IPCRR
Status: Recruiting | Type: Observational
Sponsor: Pachyonychia Congenita Project (Other)
Responsible Party: Sponsor
Other Study IDs: 20040468
Record Dates: First submitted 2014-12-12; First posted 2014-12-22 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Pachyonychia Congenita
Keywords: Nail Dystrophy; Plantar Keratoderma; Palmar Keratoderma; Leukokeratosis; Cysts; Pain; KRT17; KRT16; KRT6A; KRT6B; KRT6C
MeSH Terms: conditions — Pachyonychia Congenita; Leukoplakia; Cysts; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
International Pachyonychia Congenita Research Registry (IPCRR) is a patient registry for those suffering from Pachyonychia Congenita (PC). PC is an ultra-rare extremely painful skin disorder that causes painful blisters and callus on feet and sometimes hands, thickened nails, cysts and other features. The IPCRR consists of a questionnaire, patient photos, optional physician notes from telephone consultation to validate questionnaire and free genetic testing.

DETAILED DESCRIPTION:
HOW TO PARTICIPATE IN IPCRR

Step One: The IPCRR forms are available online at http://www.pachyonychia.org/patient-registry/. The Consent Form protects your privacy and the Questionnaire gathers important details that distinguish PC from other conditions and helps to identify specific characteristics of each type of PC. You may stop and start as often as needed before completing the forms. If you are not certain about an answer, you may skip that question.

Step Two: Take photos as shown in the Questionnaire sample photo page. You can upload the images online with the Questionnaire. If you prefer, you may email the photos. Photos of your PC are very important. Note: If you do not have access to a computer and wish to have the IPCRR forms mailed, please contact PC Project.

Step Three: When your Consent Form, Questionnaire, and Photos are received by PC Project, we will have an intake call with you to review your information and to discuss the next steps.

Step Four: If referred for genetic testing, you will then be sent the special saliva test kit (no travel required). Usually, only saliva is needed and from only one family member. The sample is collected by spitting into the vial in the kit and then mailing it in the envelope provided. Genetic testing is complex and time-consuming - it is not like a sugar test or pregnancy test, and can take many months to be completed, but the testing begins as soon as your sample arrives.

When the confirming results are received, a full genetic testing report is provided to you with precise information and suggestions specific to your condition. You may find the report very valuable with physicians or other medical providers as well as for school personnel, employers, disability hearings, or other special needs. All information is held confidentially by PC Project and the research is reported anonymously. There is no cost to you for any of these tests or assistance from PC Project. You may also request additional consultations as needed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Pachyonychia Congenita or similar disorder

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All persons with PC in all countries are being invited to register. It is not known how many persons have PC although it is known to be a very rare disease.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2004-04; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Describing patterns and traits of Pachyonychia Congenita | Once a year

CONTACTS AND LOCATIONS:
Overall Officials: C. David Hansen, MD, Principal Investigator — Pachyonychia Congenita Project
Locations (1):
- Pachyonychia Congenita Project, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Wilson NJ, O'Toole EA, Milstone LM, Hansen CD, Shepherd AA, Al-Asadi E, Schwartz ME, McLean WH, Sprecher E, Smith FJ. The molecular genetic analysis of the expanding pachyonychia congenita case collection. Br J Dermatol. 2014 Aug;171(2):343-55. doi: 10.1111/bjd.12958. Epub 2014 Aug 6. PMID 24611874
- [Background] Shah S, Boen M, Kenner-Bell B, Schwartz M, Rademaker A, Paller AS. Pachyonychia congenita in pediatric patients: natural history, features, and impact. JAMA Dermatol. 2014 Feb;150(2):146-53. doi: 10.1001/jamadermatol.2013.6448. PMID 24132595
- [Result] McLean WH, Hansen CD, Eliason MJ, Smith FJ. The phenotypic and molecular genetic features of pachyonychia congenita. J Invest Dermatol. 2011 May;131(5):1015-7. doi: 10.1038/jid.2011.59. Epub 2011 Mar 24. PMID 21430705
- [Result] Eliason MJ, Leachman SA, Feng BJ, Schwartz ME, Hansen CD. A review of the clinical phenotype of 254 patients with genetically confirmed pachyonychia congenita. J Am Acad Dermatol. 2012 Oct;67(4):680-6. doi: 10.1016/j.jaad.2011.12.009. Epub 2012 Jan 20. PMID 22264670
- See also: Pachyonychia Congenita Project Website — http://www.pachyonychia.org
- See also: Link to IPCRR information and forms — http://www.pachyonychia.org/patient-registry/
- See also: Link to data/graphs from IPCRR — http://www.pachyonychia.org/pc-data/
- See also: Link to Published Research Articles on PC — http://www.pachyonychia.org/research-articles/